CLINICAL TRIAL: NCT01709084
Title: A Phase 3b, Randomized, Open-label Clinical Study to Demonstrate Non-inferiority in Virologic Response Rates of HIV-1 RNA Suppression <400 Copies/mL of TDF/FTC/RPV Versus TDF/FTC/EFV in First-line Antiretroviral NNRTI-based Suppressed Patients. Switching At Low HIV-1 RNA Into Fixed Dose Combinations (SALIF)
Brief Title: A Clinical Trial Comparing the Efficacy of Tenofovir Disoproxil Fumarate/Emtricitabine/Rilpivirine (TDF/FTC/RPV) Versus TDF/FTC/Efavirenz (TDF/FTC/EFV) in Patients With Undetectable Plasma HIV-1 RNA on Current First-line Treatment
Acronym: SALIF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100875; TMC278IFD3002 (Other: Janssen-Cilag International NV)
Record Dates: First submitted 2012-10-16; First posted 2012-10-17 (Estimated); Results first posted 2017-01-05 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Human Immunodeficiency Virus-type 1 Infection
Keywords: Human immunodeficiency virus-type 1 infection; HIV-1; Infectious diseases; Ribonucleic acid; RNA; Tenofovir disoproxil fumarate; Emtricitabine; Rilpivirine; Efavirenz; Edurant; TMC278; R278474; Fixed dose combination
MeSH Terms: conditions — Communicable Diseases | interventions — Rilpivirine; efavirenz; Tenofovir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Patients will receive fixed dose combination (FDC) tablet of tenofovir disoproxil fumarate/emtricitabine/rilpivirine with a meal, until Week 48.
  Interventions: Drug: Rilpivirine; Drug: Tenofovir disoproxil fumarate; Drug: Emtricitabine
- Group 2 (Active Comparator): Patients will receive FDC tablet of tenofovir disoproxil fumarate/emtricitabine /efavirenz on an empty stomach at bedtime, until Week 48.
  Interventions: Drug: Efavirenz; Drug: Tenofovir disoproxil fumarate; Drug: Emtricitabine

INTERVENTIONS:
Drug: Rilpivirine — Type=exact number, unit=mg, number=25, form=tablet, route=oral. Rilpivirine will be administered in a fixed dose combination along with tenofovir disoproxil fumarate and emtricitabine, as a single dose tablet.
  Other Names: EDURANT
  Arms: Group 1
Drug: Efavirenz — Type=exact number, unit=mg, number=600, form=tablet, route=oral. Efavirenz will be administered in a fixed dose combination along with tenofovir disoproxil fumarate and emtricitabine, as a single dose tablet.
  Arms: Group 2
Drug: Tenofovir disoproxil fumarate — Type=exact number, unit=mg, number=300, form=tablet, route=oral. Tenofovir disoproxil fumarate will be administered in a fixed dose combination along with rilpivirine and emtricitabine in Group 1, and along with efavirenz and emtricitabine in Group 2.
Drug: Emtricitabine — Type=exact number, unit=mg, number=200, form=tablet, route=oral. Emtricitabine will be administered in a fixed dose combination along with rilpivirine and tenofovir disoproxil fumarate in Group 1, and along with efavirenz and tenofovir disoproxil fumarate in Group 2.

SUMMARY:
The purpose of this study is to demonstrate noninferiority (a new treatment is equivalent to standard treatment) in terms of the percentage of patients who have plasma human immunodeficiency virus-type 1 (HIV-1) ribonucleic acid (RNA) levels less than 400 copies per mL after 48 weeks of randomized treatment with tenofovir disoproxil fumarate/emtricitabine/rilpivirine (TDF/FTC/RPV) versus TDF/FTC/efavirenz (TDF/FTC/EFV).

DETAILED DESCRIPTION:
This is a 48-week, multicenter (study conducted at multiple sites), multinational (conducted at different countries), open-label (all people know the identity of the intervention), randomized (the study medication is assigned by chance) study to assess whether tenofovir disoproxil fumarate/emtricitabine/rilpivirine (TDF/FTC/RPV) shows noninferior response rates of human immunodeficiency virus-type 1 (HIV-1) ribonucleic acid (RNA) suppression less than 400 copies per mL, compared with TDF/FTC/efavirenz (TDF/FTC/EFV). The study consists of 3 phases including, the screening phase (of 6 weeks), treatment phase (of 48 weeks), and follow up phase (of 30 to 35 days after the last dose of study medication). During the 48 weeks treatment phase, patients currently with HIV-1 RNA suppression less than 50 copies per mL on their first-line antiretroviral regimen, will be randomized in a 1:1 ratio, in 2 groups, ie, Group 1 (treatment group) and Group 2 (control group). Both these groups will receive a fixed dose combination (FDC) regimen (ie, FDC tablet: one tablet per day) of either TDF/FTC/RPV in Group 1 or TDF/FTC/EFV in Group 2. Patients will return for study visits at Week 4, 12, 24, 36, and 48 during the treatment period, and then every 24 weeks thereafter during the extended treatment period until the last patient has his or her Week 48 (or treatment discontinuation) visit. Safety evaluations for adverse events, clinical laboratory (central and local) tests, electrocardiogram, vital signs, and physical examination will be performed throughout the study. The treatment duration for each patient will be expected to be between 48 and 108 weeks.

ELIGIBILITY:
Inclusion Criteria:

Documented human immunodeficiency virus-type 1 (HIV-1) infection Patients who have been receiving first line highly active antiretroviral therapy (HAART) for at least 1 year before the screening visit Patients who have been taking the same ARV combination for at least 8 weeks before the screening visit and are expected to continue on this regimen throughout the screening period.

Patients who prefer to change the current HAART regimen for reasons of simplification and/or toxicity of nucleoside/nucleotide reverse transcriptase inhibitor (N[t]RTI) Plasma HIV-1 RNA less than 50 copies per mL and CD4+ cell count higher than 200 per mm3 at the screening visit Agrees to protocol-defined use of effective contraception

Exclusion Criteria:

History of virologic failure (2 consecutive plasma HIV-1 ribonucleic acid (RNA) more than or equal to 400 copies per mL) while on previous or current ART History of immunologic failure (2 consecutive CD4+ cell counts during HAART treatment falling below the pre-HAART level) History of any primary N[t]RTI or NNRTI mutations Has a previously documented HIV-2 infection Significantly decreased hepatic function or hepatic insufficiency or diagnosed with acute clinical viral hepatitis Diagnosed with Mycobacterium tuberculosis infection Severe laboratory abnormalities Creatinine clearance less than 50 mL per minute Addicted to drug, including alcohol or recreational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2013-10-02 (Actual); Primary Completion 2015-10-22 (Actual); Study Completion 2020-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (18):
- Cameroon (2):
  - Douala
  - Yaoundé
- Kenya (4):
  - Eldoret
  - Kangemi, Nairobi
  - Nairobi
  - Nyanza
- Senegal (2):
  - Dakar
  - Pikine
- South Africa (5):
  - Bloemfontein
  - Johannesburg
  - Soweto
  - Wentworth, Durban
  - Westville, KwaZulu
- Thailand (3):
  - Amphur Mueang Nonthaburi
  - Bangkok
  - Chiang Mai
- Uganda (2):
  - Entebbe
  - Kampala

RESULTS

PARTICIPANT FLOW:
Groups:
- TDF/FTC/RPV: Participants received Film-coated fixed dose combination (FDC) tablet containing 300 milligram (mg) Tenofovir disoproxil fumarate (TDF), 200 mg Emtricitabine (FTC) and 25 mg Rilpivirine (RPV) with a meal, until Week 48.
- TDF/FTC/EFV: Participants received Film-coated fixed dose combination (FDC) tablet containing 300 milligram (mg) Tenofovir disoproxil fumarate (TDF), 200 mg Emtricitabine (FTC) and 600 mg Efavirenz (EFV) on an empty stomach at bedtime, until Week 48.
Period: Overall Study
Arm/Group | TDF/FTC/RPV | TDF/FTC/EFV
Started | 213 | 213
Treated | 213 | 211
Completed | 197 | 198
Not Completed | 16 | 15
Not completed — Lost to Follow-up | 4 | 7
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 5 | 0
Not completed — Other | 5 | 3
Not completed — Participant Reached a Virologic Endpoint | 0 | 1
Not completed — Not Treated | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TDF/FTC/RPV | TDF/FTC/EFV | Total
Number analyzed (Participants) | 213 | 211 | 424
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (8) | 40.6 (8.7) | 40.6 (8.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 134 | 271
  Male | 76 | 77 | 153
Region of Enrollment [Number; unit: participants]
  CAMEROON | 16 | 13 | 29
  KENYA | 36 | 37 | 73
  SENEGAL | 17 | 8 | 25
  SOUTH AFRICA | 33 | 30 | 63
  THAILAND | 51 | 58 | 109
  UGANDA | 60 | 65 | 125

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma Human Immunodeficiency Virus - Type 1 Ribonucleic Acid (HIV-1 RNA) Levels Less Than (<) 400 Copies Per Milliliter (Copies/mL) at Week 48
Description: Percentage of Participants with viral load (plasma HIV-1 RNA levels) less than 400 copies per mL at Week 48, obtained by the modified Food and Drug Administration (FDA) Snapshot method.
Time Frame: Week 48
Population: The intent-to-treat (ITT) population included all participants who were randomized and who had taken at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | TDF/FTC/RPV | TDF/FTC/EFV
Number analyzed (Participants) | 213 | 211
Percentage of Participants | 93.9 [lower limit -6.44] | 96.2

2. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Levels < 50 Copies/mL at Week 48
Description: Percentage of Participants with plasma HIV-1 RNA <50 copies/mL, obtained by the modified Food and Drug Administration (FDA) Snapshot method.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | TDF/FTC/RPV | TDF/FTC/EFV
Number analyzed (Participants) | 213 | 211
Percentage of Participants | 93.9 | 96.2

3. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Levels More Than or Equal to (>=) 400 Copies/mL at Week 48 Based on Time to Loss of Virologic Response (TLOVR) [Non-virologic Failure Censored] Imputation Method.
Description: Percentage of participants with plasma HIV-1 RNA levels analysed based on time to loss of virologic response (TLOVR) imputation method which is defined as confirmed plasma HIV-1 RNA >=400 copies/mL, excluding participants who discontinued the study with HIV-1 RNA suppression <400 copies/mL.
Time Frame: Week 48
Population: The intent-to-treat (ITT) population included all participants who were randomized and who had taken at least 1 dose of study drug. Here, N (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | TDF/FTC/RPV | TDF/FTC/EFV
Number analyzed (Participants) | 201 | 205
Percentage of Participants | 0.5 | 0.5

4. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Levels >= 50 Copies Per Milliliter (Copies/mL) at Week 48 Based on Time to Loss of Virologic Response (TLOVR) [Non-virologic Failure Censored] Imputation Method.
Description: Percentage of participants with plasma HIV-1 RNA levels analysed based on TLOVR imputation method which is defined as confirmed plasma HIV-1 RNA >=50 copies/mL, excluding participants who discontinued the study with HIV-1 RNA suppression <50 copies/mL.
Time Frame: Week 48
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | TDF/FTC/RPV | TDF/FTC/EFV
Number analyzed (Participants) | 201 | 205
Percentage of Participants | 1.5 | 1.0

5. Secondary Outcome: Percentage of Participant With Treatment Adherence Based on Tablet Count
Description: In both treatment groups adherence rates assessed by tablet count, the majority of participants had an adherence of >95% (97% and 98% in RPV and EFV treated treatment groups respectively).
Time Frame: Up to 48 Weeks
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | TDF/FTC/RPV | TDF/FTC/EFV
Number analyzed (Participants) | 207 | 206
Percentage of Participants | 97.2 (1.981) | 97.6 (1.649)

6. Secondary Outcome: Number of Participants With Treatment-Emergent Nucleoside Reverse Transcriptase Inhibitor (N[t]RTI) or Nucleoside/Nucleotide Reverse Transcriptase Inhibitor (NNRTI) Mutations
Description: To compare the loss of treatment options, the number of participants with treatment-emergent N[t]RTI or NNRTI mutations, as defined by IAS-USA (2014), after virologic failure were compared between the treatment groups.
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | TDF/FTC/RPV | TDF/FTC/EFV
Number analyzed (Participants) | 213 | 211
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | TDF/FTC/RPV | TDF/FTC/EFV
Serious Adverse Events (participants affected / at risk) | 16/213 | 11/211
Other Adverse Events (participants affected / at risk) | 128/213 | 137/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TDF/FTC/RPV (N=213) | TDF/FTC/EFV (N=211)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0
Gastrointestinal Inflammation (Gastrointestinal disorders) | 0 | 1
Food Allergy (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Neurocysticercosis (Infections and infestations) | 1 | 0
Neurosyphilis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 | 1
Adenomyosis (Reproductive system and breast disorders) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1
Uterine Haemorrhage (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TDF/FTC/RPV (N=213) | TDF/FTC/EFV (N=211)
Neutropenia (Blood and lymphatic system disorders) | 8 | 12
Vertigo (Ear and labyrinth disorders) | 11 | 19
Diarrhoea (Gastrointestinal disorders) | 8 | 11
Malaria (Infections and infestations) | 10 | 22
Upper Respiratory Tract Infection (Infections and infestations) | 63 | 59
Urinary Tract Infection (Infections and infestations) | 29 | 28
Amylase Increased (Investigations) | 14 | 5
Blood Pressure Increased (Investigations) | 13 | 9
Increased Appetite (Metabolism and nutrition disorders) | 11 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 15
Back Pain (Musculoskeletal and connective tissue disorders) | 20 | 14
Dizziness (Nervous system disorders) | 7 | 14
Headache (Nervous system disorders) | 38 | 29
Somnolence (Nervous system disorders) | 11 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 10
Hypertension (Vascular disorders) | 5 | 13

LIMITATIONS AND CAVEATS:
It was an open label switch study with a significant number of patients (55%) on the Efavirenz (EFV) arm who did not switch their Nucleoside/Nucleotide Reverse Transcriptase Inhibitor (NNRTI) unlike in the Rilpivirine (RPV) arm where 100% switched.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.